CLINICAL TRIAL: NCT03946488
Title: Évaluation Des modalités Optimales de Pilotage et de l'Impact Sur Les capacités de préhension d'Une Stimulation électrique Fonctionnelle Des Muscles Extenseurs Des Doigts Chez le Patient hémiplégique en Phase Chronique
Brief Title: Functional Impact of a Closed-loop Controlled Grasping Neuroprosthesis in Post-stroke Patients (PREHENSTROKE)
Acronym: PREHENSTROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LOCAL/2018/DG-01; 2018-A02144-51 (Other: ANSM)
Record Dates: First submitted 2019-04-24; First posted 2019-05-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2021-07

CONDITIONS: Stroke
Keywords: Hand function restoration; Prehension; Closed-loop controlled neuroprosthesis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inactive neuroprosthesis (No Intervention)
- Active neuroprosthesis (Experimental)
  Interventions: Device: Functional electrical stimulation

INTERVENTIONS:
Device: Functional electrical stimulation — Functional electrical stimulation of finger's muscles in order to open the hand
  Arms: Active neuroprosthesis

SUMMARY:
Stroke is the leading cause of disability in adults. The improvement of the grasp abilities remains a challenge in the 50% of post-stroke subjects who have not recovered functional grasping due to paralysis of the finger's muscles (lack of active opening of the hand).

The use of functional electrical stimulation of the prehension muscles in order to restore grasp abilities, called grasp neuroprosthesis (GP), remained confidential in post-stroke subjects while their development was important in tetraplegic subjects. GP can provide a correct hand opening with significant functional gain, but one of the major issues corresponds to the control modalities that are not adapted to the specific impairments of post-stroke subjects.

This project proposes to assess the functional contribution of an innovative autopilot closed-loop GP targeting the extensor muscles of the fingers. The main hypothesis is that the use of GP will restore grasping abilities in subjects who have lost this ability due to post-stroke paralysis.

The main objective is to assess the impact of using an autopilot closed-loop GP on the ability to perform a standardized task of grasping, moving and releasing either a glass (palmar grasp) or a spoon (key pinch), compared to the absence of GP use.

The secondary objectives of the study are: (1) to assess the impact of the GP on unimanual grasp; (2) to assess which are the preferential modes of control; (3) to assess the psycho-social impacts of GP, and (4) to assess the subject's satisfaction and tolerance to the characteristics and use of GP.

The investigators plan to include 20 post-stroke hemiplegic subjects over a period of 9 months as part of a prospective, monocentric, multi-crossover, blinded evaluation study. Subjects will have active finger extension deficit secondary to stroke, with preservation of proximal movements. Each subject will be his own control (self-pairing).

Each subject will be evaluated three times, the protocol adding approximately 1½ hours of daily assessment to routine care already received. The first visit will collect clinical data after informed consent collection. The second visit will allow to choose the optimal mode of control of the GP among 8 modalities. The third visit will test the functional gain provided by the use of GP, by comparing the success or failure of carrying out functional tasks with inactive and active GP.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given free and informed consent and signed the consent;
* The patient must be an affiliate or a beneficiary of a health insurance plan;
* The patient is hospitalized as part of routine care and available for at least 3 consecutive days of follow-up during hospitalization;
* Motor deficiency of the upper limb due to a hemorrhagic or ischemic stroke;
* Stroke more than one months old;
* Inability to perform an active extension of the long fingers (opening of the hand) to voluntarily seize an empty glass with a palmar grip (grasping task in the ARAT scale), while the subject can hold the previously placed glass passively in the hand; and / or
* Inability to perform an active thumb extension to voluntarily grasp the handle of a tablespoon (flat, like a key) with a pulpo-lateral thumb-index or key-grip (grasping task in the Wolf Motor Function Scale Test), while the subject can hold the spoon previously placed passively between thumb and index;
* Ability to sit on a chair for at least 2 hours.

Exclusion Criteria:

* The subject participates in another interventional study;
* The subject is in an exclusion period determined by a previous study;
* The subject is under the protection of justice, guardianship or curatorship;
* The subject refuses to sign or give consent;
* It is not possible to give the subject enlightened information.
* The patient is pregnant, parturient, or breastfeeding;
* Patient with pacemaker;
* Unstable epilepsy;
* Unstable cardiovascular pathology (coronary heart disease, major hypertension, heart failure);
* Dermatological problems counter-indicating the application of surface electrodes;
* Musculotendinous retractions or joint stiffness of the fingers and wrist preventing passive opening of the hand sufficient to perform the functional tasks evaluated;
* Active elbow extension limited to not reaching the ipsilateral knee, the subject sitting (limitation of the approach);
* Upper limb pain limiting movements;
* Major sensory disorders corresponding to a score of the Modified Erasmus Nottingham Sensory Assessment English version of the upper limb <10/44;
* Severe aphasia with aphasia severity scale of the Boston Diagnostic Severity Aphasia Examination <= 3, indicating that there may be a clear decrease in verbal fluency or ease and speed of understanding, with no significant limitation expression or communication;
* Unilateral spatial negligence highlighted with the bell test if the difference between omissions in the left and right fields is greater than or equal to 6;
* Common extensor digitorum muscle and / or extensor thumb muscle non-stimulable with the neuroprosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Rate of success of the main functional task | Third day
  The main functional task consist of grasping, moving and releasing either a glass (palmar grasp) or a spoon (key grip): the task (palmar grasp or key grip) preferred by the patient will be chosen.
  The assessment will consist of 24 trials with the active or inactive neuroprosthesis (12 activated and 12 inactivated), the order of the trials with / without neuroprosthesis being randomized in blocks of at least three trials. In order to limit the fatigue potentially induced by the repetition of stimulations, a pause between each trial will be respected if necessary. The maximum time allowed for the completion of each test will be 1 minute.
  A success corresponds to a complete completion of the functional task in at least 2/3 of the trials (i.e. 8/12 trials) with the activated neuroprosthesis. The success / failure score will be assessed secondarily from video recordings by a blind evaluator of the activation or not of the neuroprosthesis.

SECONDARY OUTCOMES:
Rate of success of the secondary functional task | Third day
  The secondary functional task will be the one that will not be retained as a main task (primary outcome), and consist of grasping, moving and releasing either a glass (palmar grasp) or a spoon (key grip).
  The assessment will consist of 24 trials with the active or inactive neuroprosthesis (12 activated and 12 inactivated), the order of the trials with / without neuroprosthesis being randomized in blocks of at least three trials. In order to limit the fatigue potentially induced by the repetition of stimulations, a pause between each trial will be respected if necessary. The maximum time allowed for the completion of each test will be 1 minute.
  A success corresponds to a complete completion of the functional task in at least 2/3 of the trials (i.e. 8/12 trials) with the activated neuroprosthesis. The success / failure score will be assessed secondarily from video recordings by a blind evaluator of the activation or not of the neuroprosthesis.
Comparison of the Action Research Arm Test (ARAT) performed with the inactivated (first day) and activated (day three) neuroprosthesis | First and third day
  The ARAT assess different unimanual modes of prehension. The score is between 0 (the worst) and 57 (the best). The cotation will be performed secondarily from videos by a blind evaluator.
Psychosocial Impact of Assistive Devices (PIADS) questionnaire | Third day
  The PIADS assess the psychosocial impact of the use of the neuroprosthesis in the life of the person. It is composed of 3 subscales (competence, adaptability and self-esteem), each rated between -3 (worst) and +3 (best).
Subscale "Device" from the questionnaire Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | Third day
  The subscale Device of the QUEST assess the satisfaction and tolerance with respect to the characteristics and use of the neuroprosthesis. The score is between 0 (the worst) and 5 the best).

CONTACTS AND LOCATIONS:
Overall Officials: Christine Azevedo, PhD, Study Chair — Institut National de Recherche en Informatique et en Automatique; Jérôme Froger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (2):
- France (2):
  - CHU de Nîmes, Nîmes
  - CHU de TOULOUSE, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Le Guillou R, Froger J, Morin M, Couderc M, Cormier C, Azevedo-Coste C, Gasq D. Specifications and functional impact of a self-triggered grasp neuroprosthesis developed to restore prehension in hemiparetic post-stroke subjects. Biomed Eng Online. 2024 Dec 21;23(1):129. doi: 10.1186/s12938-024-01323-y. PMID 39709421